CLINICAL TRIAL: NCT06889155
Title: Comparative Study Between Oxytocin Infusion Before and After Placental Delivery on Blood Loss During and After Cesarean Delivery in Low Risk Women.
Brief Title: Comparative Study Between Oxytocin Infusion Before and After Placental Delivery on Blood Loss During and After Cesarean Delivery .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 110
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Intraoperative Blood Loss
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin before placental delivery (Active Comparator): oxytocin infusion before placental delivery just after cord clamping 10 IU of oxytocin (Syntocinon, Novartis, Basel, Switzerland) were diluted in 500 mL of normal saline and administered through intravenous infusion over 30 minutes.
  Interventions: Drug: Oxytocin
- oxytocin after placental delivery (Active Comparator): oxytocin infusion after placental delivery 10 IU of oxytocin (Syntocinon, Novartis, Basel, Switzerland) were diluted in 500 mL of normal saline and administered through intravenous infusion over 30 minutes.
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — 10 IU of oxytocin (Syntocinon, Novartis, Basel, Switzerland) were diluted in 500 mL of normal saline and administered through intravenous infusion over 30 minutes.

SUMMARY:
Participants were randomized using computer-generated random numbers into 2 groups. Group I included 32 women who received oxytocin infusion before placental delivery just after cord clamping and group II included 32 women who received oxytocin infusion after placental delivery. In both groups 10 IU of oxytocin (Syntocinon, Novartis, Basel, Switzerland) were diluted in 500 mL of normal saline and administered through intravenous infusion over 30 minutes.

DETAILED DESCRIPTION:
Participants were randomized using computer-generated random numbers into 2 groups. Group I included 32 women who received oxytocin infusion before placental delivery just after cord clamping and group II included 32 women who received oxytocin infusion after placental delivery. In both groups 10 IU of oxytocin (Syntocinon, Novartis, Basel, Switzerland) were diluted in 500 mL of normal saline and administered through intravenous infusion over 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 40 years
* singleton full term pregnancy.
* Candidate for elective cesarean delivery under spinal anaesthesia

Exclusion Criteria:

* women at high risk for intraoperative bleeding as those with placenta previa or other placental abnormalities
* women with bleeding or coagulation disorders.
* Medical disorder associating pregnancy as preeclampsia or diabetes
* Allergy or contraindications to oxytocin
* Fetal macrosomia, or congenital anomalies
* Polyhydramnios
* Uterine abnormalities as fibroids
* Women with intraoperative complications as vascular or visceral injuries

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Intraoperative blood loss | during cesarean delivery
  This was measured by weighing the surgical sponges and the suction canisters used during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Cairo University
Locations (1):
- Armed force faculty of medicine, Cairo, Egypt